CLINICAL TRIAL: NCT05106387
Title: A Noninterventional Extension Study for Patients Treated in Study R5459-RT-1944 With Vonsetamig (BCMA x CD3 Bispecific Antibody) Who Receive a Kidney Transplant
Brief Title: An Observational Extension Study for Adult Patients Treated in Study R5459-RT-1944 Who Receive a Kidney Transplant
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R5459-RT-1956
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonsetamig in study R5459-RT-1944: Received a kidney transplant and were administered vonsetamig in study R5459-RT-1944 [NCT05092347].
  Interventions: Drug: Noninterventional

INTERVENTIONS:
Drug: Noninterventional — No investigational treatment will be given in this noninterventional extension study
  Other Names: REGN5459

SUMMARY:
The main purpose of this study is to continue to see how vonsetamig works in the body and to monitor the outcomes after kidney transplant for participants previously treated in the R5459-RT-1944 study (NCT05092347).

No study drug will be given during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Received at least 1 dose of treatment with vonsetamig in study R5459-RT-1944 [NCT05092347].
2. Received after acceptable crossmatching, a kidney transplant while enrolled in study R5459-RT-1944
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide informed consent signed by study patient or legally acceptable representative

Exclusion Criteria:

1.There are no exclusion criteria for this study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to collect safety and outcomes data in patients aged 18 through 70 years who receive a kidney transplant and were administered vosentamig in study R5459-RT-1944 [NCT05092347].
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 12 months post-kidney transplant
Incidence of Serious Adverse Events | Up to 12 months post-kidney transplant

SECONDARY OUTCOMES:
Incidence of biopsy-proven kidney allograft rejection | Up to 12 Months
  Responsiveness to therapy by 12 months of each of the following types of biopsy-proven kidney allograft rejection according to Banff classification:
  * Active antibody-mediated rejection (AMR) (Category 2)
  * Chronic active AMR (Category 2)
  * Acute t-cell-mediated rejection (TCMR) (Category 4)
  * Chronic active TCMR (Category 4)
Time to diagnosis of biopsy-proven kidney allograft rejection | Up to 12 Months
  Responsiveness to therapy by 12 months of each of the following types of biopsy-proven kidney allograft rejection according to Banff classification:
  * Active antibody-mediated rejection (AMR) (Category 2)
  * Chronic active AMR (Category 2)
  * Acute t-cell-mediated rejection (TCMR) (Category 4)
  * Chronic active TCMR (Category 4)
Responsiveness to therapy by 12 months of biopsy-proven kidney allograft rejection | Up to 12 Months
  Responsiveness to therapy by 12 months of each of the following types of biopsy-proven kidney allograft rejection according to Banff classification:
  * Active antibody-mediated rejection (AMR) (Category 2)
  * Chronic active AMR (Category 2)
  * Acute t-cell-mediated rejection (TCMR) (Category 4)
  * Chronic active TCMR (Category 4)
Incidence of graft loss | Up to 12 Months
  Incidence of graft loss (defined as becoming dialysis-dependent) by 12 months
Time to graft loss | Up to 12 Months
  Time to graft loss (defined as becoming dialysis-dependent) by 12 months
Change in estimated glomerular filtration rate (eGFR) over time | Up to 12 Months
Incidence of delayed graft function | Up to Day 7
  Incidence of delayed graft function (defined as the use of dialysis within 7 days posttransplant)
Percent Change in anti-HLA alloantibodies | Up to 12 months
  Percent Change in anti-HLA alloantibodies (SAB assay) compared with pretransplant levels at 2, 3, 6, and 12 months, and at the time of suspected clinical episodes of allograft rejection
Mean Fluorescence Intensity Change in anti-HLA alloantibodies | Up to 12 months
  Mean Fluorescence Intensity (MFI) Change in anti-HLA alloantibodies (SAB assay) compared with pretransplant levels at 2, 3, 6, and 12 months, and at the time of suspected clinical episodes of allograft rejection
Change in Calculated panel-reactive antibody (cPRA) over time | Up to 12 Months
Percent Change in donor-specific anti-HLA alloantibodies | Up to 12 Months
  Percent Change in donor-specific anti-HLA alloantibodies compared with recipient pre-transplant anti-HLA alloantibody levels
Mean Fluorescence Intensity Change in donor-specific anti-HLA alloantibodies | Up to 12 Months
  Mean Fluorescence Intensity Change in donor-specific anti-HLA alloantibodies compared with recipient pre-transplant anti-HLA alloantibody levels
Incidence of de novo anti-HLA alloantibody development | Up to 12 Months
  Cumulative incidence of de novo anti-HLA alloantibody development by SAB assay by 12 months
Serum Concentrations of Ig classes (IgG, IgA, and IgM) over time | Up to 12 Months
Percent change from baseline of circulating serum concentrations of Ig classes | Up to 12 Months
  Percent change from baseline of circulating serum concentrations of Ig classes (IgG, IgA, and IgM)
Serum Concentration of vonsetamig | Up to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - Connie Frank Transplant Center at UCSF, San Francisco, California
  - Yale University of Medicine, New Haven, Connecticut
  - Comprehensive Transplant Center, Chicago, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - New York University Langone Health, New York, New York
  - Penn Transplant Institute, Philadelphia, Pennsylvania